CLINICAL TRIAL: NCT04619849
Title: Electrophysiological Changes in the Median Nerve in the Presence and Absence of the Palmaris Longus
Brief Title: Electrophysiological Changes Based on the Palmaris Longus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gizem ergezen, Gizem Ergezen, MSc, Physiotherapist, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10840098-722.02-E.342196
Record Dates: First submitted 2020-11-03; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Palmaris Longus Muscle, Absence of; Carpal Tunnel Syndrome; EMG Syndrome
Keywords: carpal tunnel syndrome; palmaris longus; median nerve; carpal tunnel
MeSH Terms: conditions — Carpal Tunnel Syndrome; Beckwith-Wiedemann Syndrome; Median Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- palmaris longus and carpal tunnel (Experimental): EMG measurements of median and ulnar nerves will be made in patients with palmaris longus muscle.
  Interventions: Diagnostic Test: EMG; Diagnostic Test: Palmaris Longus Test

INTERVENTIONS:
Diagnostic Test: EMG — Electromyography (EMG) is an electrodiagnostic medicine technique for evaluating and recording the electrical activity produced by skeletal muscles.
Diagnostic Test: Palmaris Longus Test — Schaffer test will be done to understand the presence of palmaris longus. 4 different tests will be done to prove its absence.

SUMMARY:
One of the most important causes of carpal tunnel syndrome is increased pressure in the canal. With the loading of the palmaris longus at 20 degrees of wrist extension, the pressure within the canal increases more than the load exerted on other flexor tendons. Several studies have shown the association of carpal tunnel syndrome with the presence of palmaris longus. In this study, our aim is to investigate how the presence or absence of palmaris longus changes EMG measurements in the median nerve. Individuals with a diagnosis of carpal tunnel syndrome or entrapment neuropathy will be given the Schaffer test, a standardized test to test the presence of the palmaris longus muscle. The result will be noted, EMG examination will be requested and the electrophysiological properties of the median nerve will be recorded.

DETAILED DESCRIPTION:
One of the most important causes of carpal tunnel syndrome(CTS) is the pressure increase in the canal. With the loading of the palmaris longus at 20 degrees of wrist extension, the pressure within the canal increases more than the load exerted on other flexor tendons. Several studies have shown the association of carpal tunnel syndrome with the presence of palmaris longus. Our aim in this study is to investigate how the presence or absence of the palmaris longus changes the EMG measurements in the median nerve. Individuals with a diagnosis of carpal tunnel syndrome or entrapment neuropathy will be given the Schaffer test, a standardized test to test the presence of the palmaris longus muscle. The result will be noted, EMG examination will be requested, and the electrophysiological properties of the median nerve will be recorded. If the Schaffer test that detects the presence of palmaris longus is negative, 4 different tests that will prove the absence of palmaris longus will be performed by the same practitioner. These 4 tests are Thompson's test, Mishra's test I, Mishra's test II and Pushpakumar's "two-finger sign" method. Routine median nerve conduction studies are valuable in CTS. Prolonged distal latency in motor and sensory nerves can be found in most cases of CTS. If routine studies are insufficient, more sensitive methods are needed. These; Comparison of mixed latencies in the wrist recording of the sensory responses of the median and ulnar nerves with palmar stimulation, median and ulnar sensory latencies with orthodromic or antidromic recording from the 4th finger, median and ulnar motor latencies with recording from the second lumbrical and second interosseous muscle, median and radial sensory latencies with thumb recording It is based on determining the compression point by centrifugation method by performing segmental sensory nerve conduction examination.

ELIGIBILITY:
Inclusion Criteria:

* Applying to the electrophysiology laboratory for an EMG examination for entrapment neuropathy. The examination should be requested by a doctor.

Exclusion Criteria:

* Having a disease affecting the orthopedic, neurological or rheumatological skeletal and neurological system;
* Those who do physical activity so heavy that they cause muscle pain or neurological damage;
* Those who have an operation in the area to be evaluated

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-05 (Estimated); Primary Completion 2020-12-19 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Median Nerve Conduction Velocity | 1st day
  right and left median nerve conduction velocity will be assessed with EMG, (m/s)
Median Nerve Peak Latency | 1st day
  right and left median nerve peak latency will be assessed with EMG,0 (ms)

SECONDARY OUTCOMES:
Ulnar Nerve Conduction Velocity | 1st day
  right and left ulnar nerve conduction velocity will be assessed with EMG, (m/s)
Ulnar Nerve Peak Latency | 1st day
  right and left ulnar nerve peak latency will be assessed with EMG,0 (ms)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Şahin, PhD, Study Chair — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No